CLINICAL TRIAL: NCT06685523
Title: Evaluation of Fractalkine and Its Receptor in the Non-Surgical Treatment of Peri-implantitis
Brief Title: Evaluation of Fractalkine and Its Receptor in Peri-implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kubilay BARIŞ (Other)
Responsible Party: Sponsor-Investigator, Kubilay BARIŞ, Assistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KU-DHF-KB-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Peri-implantitis
Keywords: Er:YAG laser; Debridment; peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Four group:
  * Peri-implant healty
  * Mechanical curette
  * Er:YAG laser
  * Diyot laser
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group healty (No Intervention)
- Mechanical debridement group (Experimental)
  Interventions: Procedure: Subgingival debridement
- Er:YAG laser applied group (Experimental)
  Interventions: Procedure: Er:YAG laser decontamination
- Diyot laser applied group (Experimental)
  Interventions: Procedure: Diyot laser decontamination

INTERVENTIONS:
Procedure: Subgingival debridement — To be applied 1 times (0. days)
  Arms: Mechanical debridement group
Procedure: Er:YAG laser decontamination — To be applied 3 times
  Arms: Er:YAG laser applied group
Procedure: Diyot laser decontamination — To be applied 3 times
  Arms: Diyot laser applied group

SUMMARY:
In this study, mechanical debridement group, Er:YAG laser group and diode laser group will be compared in terms of reducing peri-implant sulcus depth in the treatment of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Probing depth of 4-6 mm, bone loss of at least 2 mm on X-ray and presence of inflammatory symptoms in soft tissue
* No systemic disease that may affect the outcome of the treatment
* Patients with healthy periodontium or patients with completed periodontal treatment
* Individuals at least 6 months after prosthesis loading on the implant
* Individuals who do not require further surgery for the treatment of peri-implantitis
* Implants with at least 2 mm keratised gingiva
* Individuals aged 40-60 years

Exclusion Criteria:

* Individuals undergoing radiation therapy
* Individuals who smoke and drink alcohol
* Individuals in pregnancy or lactation
* Individuals who have received antibiotic treatment in the last three months
* Individuals with parafunctional habits

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Probing depth, clinical attachment loss | sixth month
  Measurement will be made with a periodontal probe. The unit of measurement is millimetre. The primary outcome measures are interrelated.

SECONDARY OUTCOMES:
gingival index, plaque index, sulcus blood index | sixth month
  The 0,1,2,3 point system for index measurements is currently used in periodontology. These scores will be used in secondary outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Department of Periodontology, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No